

#### Consent to Act as a Research Subject

Physical Therapy for Latinos with Chronic Spine Pain

You are being asked to participate in a research study. Before you agree to volunteer, it is important that you know and understand what participation involves. It is important that you read the following information and ask questions as needed.

This study is funded by the National Institutes of Health (NIH).

<u>Investigators</u>: Katrina Monroe, PhD, PT and Sara P. Gombatto, PhD, PT; Doctor of Physical Therapy Program, School of Exercise and Nutritional Sciences, San Diego State University.

Purpose of the Study: The overall purpose of this study is to compare the effectiveness of two different physical therapy treatments for Hispanics/Latinos with chronic neck or back pain. Goal Oriented Activity for Latinos with Spine Pain (GOALS) is an 8-week program that combines 2 inperson evaluation sessions with 6 telephone or video treatment sessions with a physical therapist. Traditional physical therapy involves in-person treatment as recommended by a physical therapist at Family Health Centers of San Diego. The reasons you may want to participate in this study are that you may experience a decrease in pain and an improved understanding of how to manage your spine pain, activity levels, and posture and movement. Reasons you may not want to participate in this study are that you may be not be willing to participate in one of two randomly assigned physical therapy interventions for your neck or back pain. You may also feel uncomfortable sharing your personal health information with study staff, or you may not have time to participate in study-related assessments or treatment. It is also possible that you may experience no change or worsening of your pain or psychological distress with physical therapy treatment.

Participants: 138 people between the ages of 18-66 who are Hispanic or Latino, and have chronic neck or back pain will be invited to participate. Individuals who participate must have been referred by their doctor for physical therapy treatment of neck or low back pain that has persisted for at least 3 months and has resulted in pain on at least half the days in the past 6 months. They must also have eligible scores on health screening questionnaires. Once enrolled in the study, participants must attend at least 1 physical therapy treatment session in order to stay eligible. Individuals will be excluded from participating if they have a tumor, infection or other major medical problem affecting the neck or low back, have health problems that severely affect the ability to move, are involved in a lawsuit or compensation claim related to their pain condition, are pregnant or lactating, have plans to start any new behavioral health or psychological treatment for the neck or low back pain during the study period, have a diagnosis of a major psychological condition, are unable to provide a stable address with access to a telephone, are cohabitating with a GOALS/Metas participant, or any other reason that would not allow participation in a tele-rehabilitation intervention.

<u>Description of the Study</u>: If you are eligible and agree to participate, you will be asked to participate in 4 study assessments, and 8-weeks of treatment with either GOALS or traditional physical therapy. All assessments will be completed at the San Diego State University (SDSU) HealthLINK Center. If unable to travel to SDSU for study-related assessments, you will have the

option to complete these visits from your home by telephone or online video. All in-person physications 2023 therapy sessions will be completed either at Family Health Centers of San Diego (FHCSD) or the SDSU HealthLINK Center. Remote treatment sessions for the GOALS program will be completed in your own home by telephone or video.

Study assessments will last approximately 1 ½ - 2 hours, and will be scheduled 1-week before and 1-week, 3-months, and 6-months after completing the 8-weeks of GOALS or traditional physical therapy. You will be asked to complete questionnaires at the first assessment that ask about personal and demographic information (e.g. age, gender, etc.), medical history, medication use, cultural identity, and preferred language. All assessment visits will include additional surveys that ask about your physical activity, mood, environment, social support, activities, and pain intensity and disability. Post-treatment assessments will also ask about your perceived change and satisfaction with treatment.

For the first two assessment visits, you will be asked to wear small sensor devices that allow us to measure your physical activity (ActiGraph) and lower back posture and movement (Spine Motion Monitor) during your normal daily activities. You will only be given the Spine Motion Monitor if assessments are completed in-person since this requires research staff to place the monitor on your neck or back. After placing the Spine Motion Monitor on your neck or back, you will be asked to complete a movement assessment. This consists of various positions and movements that will be video recorded so that your physical therapist can assess your movement. You will be asked to wear the Spine Motion Monitor at home and/or work for up to two 8-hour days, and the physical activity monitor for seven 24-hour days to monitor your normal daily activities. You will also be given a brief questionnaire to track when you wear the physical activity monitor and your sleep behavior during the 7 days of physical activity monitoring. When monitoring is complete, you will return the sensors and the portable electronic device to study staff using a pre-paid postage return envelope. You may also choose to drop off the devices to study staff at a pick-up location and time you select in advance.

Participation in this study does not involve any invasive procedures. No information obtained from questionnaires, mobile sensors, or the portable electronic devices will be shared with your health care provider or anyone else other than study staff unless you provide written permission. Information from the screening questionnaires will be added to the research data collected from surveys and sensors. All research data for this study will be obtained by trained investigators.

After you complete the first assessment, you will be randomly assigned to participate in one of the two physical therapy interventions for chronic neck or low back pain. Random assignment means that you have an equal chance of participating in the GOALS program or traditional physical therapy at FHCSD. If you do not want to participate in the physical therapy intervention to which you are assigned, you may choose to withdraw from the study without penalty. If you withdraw from the study, you will be referred back to FHCSD to continue your normal course of care.

The 8-week GOALS intervention involves one 60-minute evaluation with a physical therapist, followed by 7 treatment sessions with the same therapist for approximately 45 minutes, once a week. Six of the 7 treatment sessions will be conducted in your home by telephone, with one session conducted in-person so that your physical therapist can make sure you are doing your exercises correctly. In total, for the GOALS treatment, you will be required to travel to either FHCSD or the SDSU HealthLINK Center for two in-person sessions with your physical therapist. If you are unable to travel to the clinic for in-person sessions, you will have the option to attend through a secure online video call instead. All physical therapy sessions will be audio recorded so that we can monitor what treatments you receive at each session. In the GOALS program, your

physical therapist will teach you different ways to manage your pain using therapeutic exercise? August 2023 deep breathing, balancing your activity with rest, getting support from others, being present in the moment, balancing your thinking, and creating a plan to stay healthy after you finish the program. Each week, you will create goals for doing your physical therapy exercises, walking, getting back to daily activities that are important to you, and practicing new ways to manage your pain. Your physical therapist will also teach you how to exercise and move safely so you can be more active throughout your day. You will receive exercise equipment to take home, and a booklet that has pictures and written instructions in your preferred language to help you follow along with your physical therapist at each treatment session and remember what activities to do on your own between sessions.

The traditional physical therapy program involves one 30-minute evaluation with a physical therapist at FHCSD, followed by in-person physical therapy treatment sessions as recommended by your physical therapist. All evaluation and treatment sessions will require you to travel to a FHCSD clinic to receive care. Physical therapy treatments may include therapeutic exercise, modalities (e.g. heat/ice, traction, electrical stimulation), manual therapy (e.g. spine mobilization/manipulation, soft-tissue massage, stretching), advice on how to move safely during your daily activities, or other treatments recommended by your physical therapist. Your physical therapist will determine the frequency and duration of physical therapy sessions required after your initial evaluation. If your care extends longer than 8-weeks, you will return for study assessments after completing 8-weeks of treatment, and then 3-months and 6-months of later, but you will continue to receive care as usual from your physical therapist.

What is Experimental in this Study?: In a previous study for post-surgical spine pain, a tele-rehabilitation program similar to GOALS was acceptable to patients and resulted in a clinically meaningful improvement in pain and disability. Adapting and applying this intervention for Hispanics and Latinos with chronic spine pain is the experimental component of this study.

**Risks or Discomforts**: You will be asked to provide personal information through questionnaires and wearable activity monitoring devices. There is potential for embarrassment about or other negative reactions to discussion of personal health-related behaviors and feelings. For assessments with the Spine Motion Monitor, it is possible that the adhesive used to apply the sensors can produce skin redness, irritation, discomfort on removal, or increased pain with certain movements. You may decline any individual question, measurement, or the entire assessment session at any time without penalty.

For the physical therapy intervention, you may experience increased spine pain, muscle soreness, or psychological stress associated with participation in either the GOALS program or traditional physical therapy. However, these symptoms are typical when starting a new exercise program and generally improve within 48 hours. All changes in symptoms during treatment will be monitored and addressed by your physical therapist. If at any time during the study your physical therapist determines that you require additional medical attention, they will refer you back to your primary care physician at FHCSD for care.

You may also feel uncomfortable having your conversations recorded during treatment or being recorded while completing the movement assessments. However, we will keep all audio tapes private and any information that personally identifies you will be removed. We will not share these recordings with anyone without your written consent.

Overall, both interventions are considered minimal risk, and have been shown to be effective for patients with chronic neck or back pain. You may decline any individual component or the entire

intervention at any time without penalty.

If during any portion of the study, research staff or your physical therapist determine that you demonstrate significant depression, suicidal intent or plan, you will be encouraged to seek immediate medical attention. If you are not willing to seek medical attention, research staff will be required to contact local mental health resources for guidance.

<u>Benefits</u>: You may experience a clinically meaningful decrease in pain and an improved understanding of how to manage your spine pain, activity levels, and posture and movement. It is also possible that science and society will benefit from a better understanding of the effects ofa tele-rehabilitation program for chronic spine pain in Hispanics and Latinos. However, we cannot guarantee that you will receive any direct benefits from participating in this study.

<u>Alternatives to Participation</u>: Participation in this study is voluntary and you have the alternative of not participating or withdrawing at any time without penalty. If you choose not to participate, you may resume or continue your usual course of care at FHCSD.

#### **Confidentiality/Privacy**:

All data acquired for the purposes of research will remain confidential. This research is covered by a Certificate of Confidentiality from the National Institutes of Health (NIH). This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations. Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

By agreeing to participate in this study, you are allowing study staff to access information from your electronic health record (EHR) at FHCSD. Information from the EHR that will be shared with the research team includes: dates of physical therapy referral and treatment for neck or low back pain, clinic location and number of visits attended, and type of physical therapy treatments received. All information collected from the EHR and during study visits will be coded upon study enrollment using a unique identifier before being stored on REDCap (Research Electronic Data Capture) Cloud or the SDSU HealthLINK CTHDR Health Data Analytic Portal. REDCap Cloud is a secure, password-protected, and HIPAA compliant online platform used for collecting research data. SDSU HealthLINK CTHDR Health Data Analytic Portal is a password protected HIPAA-compliant secure network server.

Study findings will be reported as group summaries, and you will not be identified by name at any time. With your additional permission (see below), de-identified data may be: 1) used by the researchers in this study or other researchers for future research, or 2) used for training purposes. De-identified data means that we will remove all information that could personally identify you from

study-related records, including audio recorded treatment sessions, prior to using using these <sup>10</sup> August <sup>2023</sup> materials for future research or training. Additionally, study-related assessment and treatment records will only be released to your health care provider or another third party with your written permission. Protected health information will be transmitted using electronic, internet, email, or facsimile devices only if appropriately encrypted and with the appropriate approvals as outlined above.

Federal regulations require that the university Institutional Review Board (IRB), Food and Drug Administration (FDA) and/or other government officials periodically review all approved and continuing projects that involve human subjects. It is possible that a representative of one of these organizations may inspect the research site and study records at any time to make sure that the study is being conducted in a safe and proper manner.

<u>Incentives to Participate</u>: You will be responsible for transportation to and from all in-person sessions conducted at FHCSD and the SDSU HealthLINK Center. Parking, snacks, and childcare (if requested) will be provided at no cost. With prior notice, transportation to and from FHCSD or the SDSU HealthLINK Center can be arranged at no cost if you have a transportation need. You may also choose to participate in these sessions through a secure video call.

You will be reimbursed with \$50 in cash for completion of outcome assessments at two of the time points (baseline and1-week post), with an additional \$50 in cash provided after the first two assessments upon return of portable monitoring devices with at least 4 valid days of activity data. You will be reimbursed with an additional \$25 in cash for completing a limited number of surveys at the 3-month and 6-month post assessments. In addition, you will receive an additional \$25 at the end of your participation if you complete all study tasks. In summary, you may earn a total of up to \$275 in cash for your participation in this study if you complete all portions of the study (8-weeks of physical therapy intervention and 4 assessments). If you choose to complete some but not all of portions of this study, you will be reimbursed for the sessions you complete.

| Study Time Point | Amount |
|------------------------------------------------|--------|
| Baseline Assessment: DorsaVi Sensor Return | \$50 |
| Baseline Assessment: Actigraph Sensor Return | \$50 |
| 1-Week Post-Assessment DorsaVi Sensor Return | \$50 |
| 1-Week Post-Assessment Actigraph Sensor Return | \$50 |
| 3-Month Post-Assessment | \$25 |
| 6-Month Post-Assessment | \$25 |
| Bonus for completing all study time points | \$25 |
| TOTAL | \$275 |

<u>Costs/Compensation for Participation</u>: If you are assigned to receive traditional physical therapy, you will be financially responsible for any co-payments billed by FHCSD that are not covered by your insurance. This is no more than the usual cost of care provided by a physical therapist at FHCSD. There are no other costs associated with participation in this study.

**Compensation for Injury**: If any complications arise as a direct result of participation in this study, we will assist you in obtaining appropriate medical attention. If you need treatment or hospitalization as a result of being in this study, you are responsible for payment of the cost for that care. If you have insurance, you may bill your insurance company. You will have to pay anycosts not covered

Approved Minimal Risk

by your insurance. San Diego State University or San Diego State University Foundation will not August 2023 pay for any care, lost wages, or provide other financial compensation.

However, if you feel you have a claim that you wish to file against the State or the Foundation, please contact Graduate and Research Affairs - SDSU Human Research Protection Program at (619) 594-6622to obtain the appropriate claim forms.

<u>Voluntary Participation</u>: Participation in this study is voluntary. Your choice of whether or notto participate will not influence your future relations with San Diego State University, San Diego State University Foundation, or Family Health Centers of San Diego. If you decide to participate, you are free to withdraw your consent and to stop your participation at any time without penalty or loss of benefits to which you are allowed.

Questions/Concerns: If you have any questions or concerns about participating in this study, please ask. If you have questions later about the research or your participation, you may contact either principal investigator, Dr. Katrina Monroe, PhD, PT (phone: 619-594-5553; email: ksmonroe@sdsu.edu) or Dr. Sara Gombatto, PhD, PT (phone: 619-594-3288; email: sgombatto@sdsu.edu). If you have any questions about your rights as a participant in this study, you may contact an IRB representative in the Division of Research Affairs at San DiegoState University (telephone: 619-594-6622; email: irb@sdsu.edu).

<u>Consent to Participate/Rights of Participant:</u> The San Diego State University Institutional Review Board has approved this consent form, as signified by the Board's stamp.

| , , | assessment and physical therapy evaluation and treatment an Diego (FHCSD) to ensure continuity of care. |
|---|---|
| (participant initials) | (date) |
| I consent to de-identified audio record related records to be used for training | lings of my physical therapy sessions and other study-<br>purposes. |
| (participant initials) | (date) |
| I consent to allow de-identified data corepository for future research. | ollected as part of this study to be placed in a data |
| (participant initials) | (date) |
| you are interested, we will contact you decide whether to participate in them | d in getting information about additional research studies. If u by phone with information about these studies and you can or not. These additional studies are separate from this study affect your ability to continue to participate in this study: |
| I consent to be contacted for future re | search opportunities as described. |
| (participant initials) | (date) |

Approved Minimal Risk

Your signature below indicates that you have read the information in this document and have Madugust 2023 chance to ask any questions you have about the study. Your signature also indicates thatyou agree to be in the study and have been told that you can change your mind and withdraw your consent to participate at any time. You have been given a copy of this consent form. You have been told that by signing this consent form you are not giving up any of your legal rights.

| Participant Name (printed) | Participant Signature | Date |
|----------------------------|-------------------------------------|------|
| | Signature of Project Representative | Date |

# Addendum to Consent to Act as a Research Subject

| GOALS/Metas researchers are reconsenting you at this time to inform you of an increase in the incentive that was approved via an amendment to this project. Please check <u>Yes</u> or <u>No</u> below indicate whether you understand you are receiving this incentive in addition to the amount you already received to better reflect the time you have dedicated to the project. | to |
|---|---|
| Yes No | |
| If you selected Yes, please initial and date below to acknowledge you agree to the additional incentive. | |
| (participant initials) (date) | |

### Addendum to Consent to Act as a Research Subject

GOALS/Metas researchers are reconsenting you at this time to inform you that additional research opportunities may be presented to you. This was approved via an amendment to this project. If you are interested, we will contact you by phone with information about these studies and you can decide whether to participate in them or not. These additional studies are separate from the GOALS/Metas study and your decisions about them will not affect your ability to continue to participate in this study.

| I consent to be contacted for future resea | arch opportunities as described above. |
|---|---|
| Yes No | |
| If you selected Yes, please initial and da<br>GOALS/Metas team about additional res | te below to acknowledge you agree to be contacted by the search studies. |
| (participant initials) | (date) |



#### Consentimiento para Actuar Como Sujeto de Investigación Terapia Física para Latinos con Dolor de Columna

Se le pide que participe en un estudió de investigación. Antes de aceptar ser voluntario, es importante que sepa y comprenda lo que implica la participación. Es importante que lea la siguiente información y haga las preguntas que necesite.

Este estudio está financiado por los Institutos Nacionales de la Salud (NIH).

<u>Investigadores</u>: Katrina Monroe, PhD, PT and Sara P. Gombatto, PhD, PT; Doctor of Physical Therapy Program, School of Exercise and Nutritional Sciences, San Diego State University.

Propósito del Estudio: El propósito general de este estudio es comparar la efectividad de dos tratamientos de fisioterapia diferentes para Hispanos/Latinos con dolor crónico de cuello o espalda. La actividad orientada a objetivos para Latinos con dolor de columna (GOALS) es un programa de 8 semanas que combina 2 sesiones de evaluación en persona con 6 sesiones de tratamiento por teléfono o video con un fisioterapeuta. La fisioterapia tradicional implica el tratamiento en persona según lo recomendado por un fisioterapeuta en Family Health Centers de San Diego. Las razones por las que puede querer participar en este estudio son que puede experimentar una disminución del dolor y una mejor comprensión de cómo manejar el dolor de la columna, los niveles de actividad, la postura y el movimiento. Es posible que no desee participar en este estudio debido a que es posible que no esté dispuesto a participar en una de las dos intervenciones de fisioterapia asignadas al azar para el dolor de cuello o espalda. También puede sentirse incómodo al compartir su información de salud personal con el personal del estudio, o puede que no tenga tiempo para participar en evaluaciones o tratamientos relacionados con el estudio. También es posible que no experimente ningún cambio o empeoramiento de su dolor o angustia psicológica con el tratamiento de fisioterapia.

**Participantes**: Se invitará a participar a 138 personas de edades entre 18 y 66 años que sean Hispanos o Latinos y que tengan dolor crónico de cuello o espalda. Las personas que participen deben haber sido referidos por su médico para el tratamiento de fisioterapia del dolor de cuello o de espalda que ha persistido durante al menos 3 meses y ha provocado dolor al menos la mitad de los días en los últimos 6 meses. También deben tener calificaciones elegibles en los cuestionarios de detección de salud. Una vez inscrito en el estudio, participantes deben asistir al menos 1 sesión de tratamiento de fisioterapia para seguir siendo elegibles. Las personas serán excluidas de participar si tienen un tumor, infección u otro problema médico importante que afecte el cuello o la espalda baja, tienen problemas de salud que afectan gravemente la capacidad de moverse, están involucrados en una demanda o reclamo de compensación relacionado con su condición de dolor, está embarazada o en período de lactancia, tiene planes de iniciar un nuevo tratamiento de salud conductual o psicológica para el dolor de cuello o lumbar durante el período de estudio, tiene un diagnóstico de una afección psicológica grave, no puede proporcionar una dirección estable con acceso a un teléfono, está actualmente viviendo con un participante del estudio GOALS/Metas, o por cualquier otro motivo que no permitiría la participación en una intervención de tele-rehabilitación.

Descripción del Estudio: Si es elegible y acepta participar, se le pedirá que participe en 4

evaluaciones del estudió, y 8 semanas de tratamiento con GOALS o fisioterapia tradicional. Todas gust 2023 las evaluaciones se completarán en el Centro HealthLINK de San Diego State University (SDSU). Si no puede viajar a SDSU para las evaluaciones relacionadas con el estudio, tendrá la opción de completar estas visitas desde su hogar por teléfono o video en línea. Todas las sesiones de fisioterapia en persona se realizarán en los Family Health Centers of San Diego (FHCSD) o en el Centro SDSU HealthLINK. Las sesiones de tratamiento a distancia para el programa GOALS se realizarán en su propia casa por teléfono o video.

Las evaluaciones del estudio durarán aproximadamente 1 ½ - 2 horas, y se programarán 1 semana antes y 1 semana, 3 meses y 6 meses después de completar las 8 semanas de GOALS o fisioterapia tradicional. Se le pedirá que complete cuestionarios en la primera evaluación que preguntan sobre información personal y demográfica (por ejemplo, edad, genero, etc.), historial médico, uso de medicamentos, identidad cultural e idioma preferido. Todas las visitas de evaluación incluirán encuestas adicionales que preguntan sobre su actividad física, estado de ánimo, ambiente, apoyo social, actividades, e intensidad del dolor y discapacidad. Las evaluaciones posteriores al tratamiento también le preguntarán sobre su cambio percibido y su satisfacción con el tratamiento.

Para las dos primeras visitas de evaluación, se le pedirá que use pequeños dispositivos sensores que nos permitan medir su actividad física (ActiGraph) y la postura y el movimiento de la espalda baja (Spine Motion Monitor) durante sus actividades diarias normales. Solo se le entregará el Monitor de movimiento de la columna vertebral (Spine Motion Monitor) si las evaluaciones se realizan en persona, ya que esto requiere que el personal de investigación coloque el monitor en su cuello o espalda. Después de colocar el monitor de movimiento de la columna vertebral en el cuello o la espalda, se le pedirá que complete una evaluación del movimiento. Consiste en varias posiciones y movimientos que se grabarán en video para que su fisioterapeuta pueda evaluar su movimiento. Se le pedirá que use el monitor de movimiento de la columna vertebral (Spine Motion Monitor) en casa y/o el trabajo hasta dos días de 8 horas, y el monitor de actividad física durante siete días de 24 horas para controlar sus actividades diarias normales. También se le entregará un breve cuestionario para rastrear cuándo usa el monitor de actividad física y su comportamiento de sueño durante los 7 días de monitoreo de actividad física. Cuando se complete el monitoreo, devolverá los sensores y el dispositivo electrónico portátil al personal del estudio utilizando un sobre de devolución prepagado. También puede optar por dejar los dispositivos para el personal del estudio en un lugar de recogida y a la hora que seleccione por adelantado.

La participación en este estudio no implica ningún procedimiento invasivo. Ninguna información obtenida de cuestionarios, sensores móviles o dispositivos electrónicos portátiles se compartirá con su proveedor de atención médica ni con ninguna otra persona que no sea el personal del estudio, a menos que proporcione un permiso por escrito. La información de los cuestionarios de selección se agregará a los datos de investigación reunidos de encuestas y sensores. Todos los datos de investigación para este estudio serán obtenidos por investigadores capacitados.

Después de completar la primera evaluación, se le asignará al azar para participar en una de las dos intervenciones de fisioterapia para el dolor crónico de cuello o espalda. La asignación aleatoria significa que tiene las mismas posibilidades de participar en el programa GOALS o en la fisioterapia tradicional en FHCSD. Si no desea participar en la intervención de fisioterapia a la que está asignado, puede optar por retirarse del estudio sin penalización. Si se retira del estudio, será referido nuevamente a FHCSD para continuar con su curso normal de cuidado.

La intervención GOALS de 8 semanas implica una evaluación de 60 minutos con un fisioterapeuta, seguida de 7 sesiones de tratamiento con el mismo terapeuta durante aproximadamente 45

minutos, una vez a la semana. Seis de las 7 sesiones de tratamiento se llevarán a cabo en sul 0 August 2023 hogar por teléfono, y una sesión se realizará en persona para que su fisioterapeuta pueda asegurarse de que está haciendo sus ejercicios correctamente. En total, para el tratamiento GOALS, se le pedirá que viaje a FHCSD o al SDSU HealthLINK Center para dos sesiones en persona con su fisioterapeuta. Si no puede viajar a la clínica para las sesiones en persona, tendrá la opción de asistir a través de una videollamada segura en línea. Todas las sesiones de fisioterapia se grabarán en audio para que podamos controlar qué tratamientos recibe en cada sesión. En el programa GOALS, su fisioterapeuta le enseñará diferentes formas de manejar su dolor mediante el ejercicio terapéutico, la respiración profunda, el equilibrio de su actividad con el descanso, el apoyo de los demás, estar presente en el momento, equilibrar su pensamiento y crear un plan para mantenerse saludable después de terminar el programa. Cada semana, creará metas para hacer sus ejercicios de fisioterapia, caminar, volver a las actividades diarias que son importantes para usted y practicar nuevas formas de controlar su dolor. Su fisioterapeuta también le enseñará cómo hacer ejercicio y moverse de manera segura para que pueda estar más activo durante el día. Recibirá equipo de ejercicio para llevar a casa, y un folleto con imágenes e instrucciones escritas en su idioma preferido para ayudarlo a seguir con su fisioterapeuta en cada sesión de tratamiento y recordar qué actividades debe hacer por su cuenta entre sesiones.

El programa de fisioterapia tradicional implica una evaluación de 30 minutos con un fisioterapeuta en FHCSD, seguida de sesiones de tratamiento de fisioterapia en persona según lo recomendado por su fisioterapeuta. Todas las sesiones de evaluación y tratamiento requerirán que viaje a una clínica de FHCSD para recibir atención. Los tratamientos de fisioterapia pueden incluir ejercicio terapéutico, modalidades (por ejemplo, calor / hielo, tracción, estimulación eléctrica), terapia manual (por ejemplo, movilización / manipulación de la columna, masaje de tejidos blandos, estiramiento), consejos sobre cómo moverse de forma segura durante sus actividades diarias, u otros tratamientos recomendados por su fisioterapeuta. Su fisioterapeuta determinará la frecuencia y duración de las sesiones de fisioterapia necesarias después de su evaluación inicial. Si su cuidado se extiende por más de 8 semanas, regresará para las evaluaciones del estudio después de completar las 8 semanas de tratamiento, y luego 3 meses y 6 meses más tarde, pero continuará recibiendo el cuidado habitual de su fisioterapeuta.

¿Qué es experimental en este estudio?: En un estudio anterior para el dolor de columna posquirúrgico, un programa de tele-rehabilitación similar a GOALS fue aceptable para los pacientes y resultó en una mejora clínicamente significativa en el dolor y la discapacidad. Adaptar y aplicar esta intervención para hispanos y latinos con dolor de columna crónico es el componente experimental de este estudio.

Riesgos o molestias: Se le pedirá que proporcione información personal a través de cuestionarios y dispositivos portátiles de monitoreo de actividad. Existe la posibilidad de vergüenza u otras reacciones negativas a la discusión de comportamientos y sentimientos personales relacionados con la salud. Para las evaluaciones con Spine Motion Monitor, es posible que el adhesivo utilizado para aplicar los sensores pueda producir enrojecimiento de la piel, irritación, malestar al retirarlo o aumento del dolor con ciertos movimientos. Puede rechazar cualquier pregunta individual, medición o la sesión de evaluación completa en cualquier momento sin penalización.

Para la intervención de fisioterapia, puede experimentar un aumento del dolor en la columna, dolor muscular o estrés psicológico asociado con la participación en el programa GOALS o en la fisioterapia tradicional. Sin embargo, estos síntomas son típicos al comenzar un nuevo programa de ejercicios y generalmente mejoran en 48 horas. Su fisioterapeuta monitoreara y abordara todos los cambios en los síntomas durante el tratamiento. Si en cualquier momento durante el estudio su fisioterapeuta

determina que necesita atención médica adicional, lo remitirán nuevamente a su médico de atención primaria en FHCSD para recibir atención.

También puede sentirse incómodo al grabar sus conversaciones durante el tratamiento o al realizar las evaluaciones de movimiento. Sin embargo, mantendremos la privacidad de todas las cintas de audio y se eliminará cualquier información que lo identifique personalmente. No compartiremos estas grabaciones con nadie sin su consentimiento por escrito.

En general, ambas intervenciones se consideran de riesgo mínimo y se ha demostrado que son efectivas para pacientes con dolor crónico de cuello o espalda. Puede rechazar cualquier componente individual o la intervención completa en cualquier momento sin penalización.

Si durante cualquier parte del estudio, el personal de investigación o su fisioterapeuta determinan que usted demuestra depresión significativa, intención o plan suicida, se le animará a buscar atención médica inmediata. Si no está dispuesto a buscar atención médica, el personal de investigación deberá comunicarse con los recursos locales de salud mental para obtener orientación.

<u>Beneficios</u>: Puede experimentar una disminución clínicamente significativa del dolor y una mejor comprensión de cómo controlar el dolor de la columna, los niveles de actividad, la postura y el movimiento. También es posible que la ciencia y la sociedad se beneficien de una mejor comprensión de los efectos de un programa de telerehabilitación para el dolor de columna crónico en hispanos y latinos. Sin embargo, no podemos garantizar que recibirá ningún beneficio directo por participar en este estudio.

<u>Alternativas a la Participación</u>: La participación en este estudio es voluntaria y tiene la alternativa de no participar o retirarse en cualquier momento sin penalización. Si elige no participar, puede reanudar o continuar su curso habitual de atención en FHCSD.

#### Confidencialidad/Privacidad:

Todos los datos adquiridos con fines de investigación serán confidenciales. Esta investigación está cubierta por un Certificado de Confidencialidad de los Institutos Nacionales de Salud (NIH). Esto significa que los investigadores no pueden divulgar ni utilizar información, documentos o muestras que puedan identificarlo en cualquier acción o juicio a menos que usted lo autorice. Tampoco pueden proporcionarlos como evidencia a menos que usted hava aceptado. Esta protección incluye procedimientos civiles, penales, administrativos, legislativos u otros procedimientos federales, estatales o locales. Un ejemplo sería una citación judicial. El Certificado NO deja de informar que exigen las leyes federales, estatales o locales. Algunos ejemplos son las leyes que exigen denunciar el abuso de niños o ancianos, algunas enfermedades transmisibles y amenazas de hacerse daño a sí mismo o a otros. El Certificado NO SE PUEDE UTILIZAR para impedir que una agencia patrocinadora del gobierno federal o estatal de los Estados Unidos verifique registros o evalúe programas. El Certificado NO detiene las divulgaciones requeridas por la Administración de Drogas y Alimentos (FDA) federal. El Certificado tampoco impide que su información se utilice para otras investigaciones si lo permiten los reglamentos federales. Los investigadores pueden divulgar información sobre usted cuando usted lo autorice. Por ejemplo, puede darles permiso para divulgar información a aseguradoras, proveedores médicos o cualquier otra persona que no esté relacionada con la investigación. El Certificado de Confidencialidad no le impide divulgar voluntariamente información sobre su participación en esta investigación. Tampoco le impide tener acceso a su propia información.

Al aceptar participar en este estudio, está permitiendo que el personal del estudio acceda a la¹º August 2023 información de su expediente médico electrónico (EHR) en FHCSD. La información del EHR que se compartirá con el equipo de investigación incluye: fechas de derivación de fisioterapia y tratamiento para el dolor de cuello o espalda, ubicación de la clínica y número de visitas asistidas, y tipo de tratamientos de fisioterapia recibidos. Su información colectada del EHR y durante sus visitas del estudio se codificará al inscribirse en el estudio utilizando un identificador único antes de almacenarse en la nube REDCap (captura de datos electrónicos de investigación) o en el Portal de Análisis de Datos de Salud SDSU HealthLINK CTHDR. REDCap Cloud es una plataforma en línea segura, protegida por contraseña y compatible con HIPAA que se utiliza para recopilar datos de investigación. El Portal de Análisis de Datos de Salud SDSU HealthLINK CTHDR es un servidor de red seguro protegido por contraseña que cumple con HIPAA.

Los resultados del estudio se informarán como resúmenes de grupo y no se le identificará por su nombre en ningún momento. Con su permiso adicional (ver más abajo), los datos no identificados pueden ser: 1) utilizados por los investigadores de este estudio u otros investigadores para investigaciones futuras, o 2) utilizados con fines de capacitación. Datos no identificados significa que eliminaremos toda la información que podría identificarlo personalmente de los registros del estudio, incluyendo sesiones de tratamiento grabadas en audio, antes de usar estos materiales para futuras investigaciones o capacitación. Además, los registros de evaluación y tratamiento relacionados con el estudio solo se divulgarán a su proveedor de atención médica u otro tercero con su permiso por escrito. La información médica protegida se transmitirá mediante dispositivos electrónicos, de Internet, correo electrónico o fax solo si está debidamente cifrada y con las aprobaciones correspondientes, como se describe anteriormente.

Las regulaciones federales requieren que la Junta de Revisión Institucional (IRB) de la universidad, la Administración de Alimentos y Medicamentos (FDA) y / u otros funcionarios gubernamentales revisen periódicamente todos los proyectos aprobados y continuos que involucran a seres humanos. Es posible que un representante de una de estas organizaciones pueda inspeccionar el sitio de investigación y los registros del estudio en cualquier momento para asegurarse de que el estudio se esté realizando de manera segura y adecuada.

Incentivos para Participar: Usted será responsable del transporte hacia y desde todas las sesiones en persona realizadas en FHCSD y el SDSU HealthLINK Center. Se proporcionará estacionamiento, refrigerios y cuidado de niños (si se solicita) sin costo alguno. Con aviso previo, el transporte desde y hacia FHCSD o el Centro HealthLINK de SDSU se puede arreglar sin costo si usted necesita transporte. También puede optar por participar en estas sesiones a través de una videollamada segura.

Se le reembolsará con \$50 por completar las evaluaciones de resultados en dos de los puntos de tiempo (línea de base y publicación de 1 semana), \$50 adicionales proporcionados después de las dos primeras evaluaciones al devolver los dispositivos portátiles con al menos 4 días válidos de datos de actividad. Se le reembolsará \$25 adicionales por completar un número limitado de encuestas en los 3 meses y 6 meses posteriores a la evaluación. Además, recibirá \$25 adicionales al final de su participación si completa todas las tareas de estudio. En resumen, puede ganar un total de hasta \$275 por su participación en este estudio si completa todas las partes del estudio (8 semanas de intervención de fisioterapia y 4 evaluaciones). Si opta por completar algunas partes de este estudio, pero no todas, se le reembolsarán las sesiones que complete.

| Partes del Estudio | Cantidad |
|----------------------------------------------------------------|----------|
| Evaluación Base: Regreso del sensor DorsaVi | \$50 |
| Evaluación Base: Regreso del sensor Actigraph | \$50 |
| Evaluación 1 semana después de completar tratamiento: Regreso | \$50 |
| del sensor DorsaVi | |
| Evaluación 1 semana después de completar tratamiento: Regreso | \$50 |
| del sensor Actigraph | |
| Evaluación de 3 mess | \$25 |
| Evaluación de 6 meses | \$25 |
| Incentivo adicional por completar todas las partes del estudio | \$25 |
| TOTAL | \$275 |

<u>Costos/Compensación por Participación:</u> Si se le asigna a recibir fisioterapia tradicional, será financieramente responsable de cualquier copago facturado por FHCSD que no esté cubierto por su seguro. Este no es más que el costo habitual de la atención brindada por un fisioterapeuta en FHCSD. No hay otros costos asociados con la participación en este estudio.

<u>Compensación por Lesiones</u>: Si surge alguna complicación como resultado directo de la participación en este estudio, lo ayudaremos a obtener la atención médica adecuada. Si necesita tratamiento u hospitalización como resultado de participar en este estudio, usted es responsable del pago del costo de esa atención. Si tiene seguro, puede facturar a su compañía de seguros. Tendrá que pagar los gastos que no cubra su seguro. San Diego State University o la Fundación de San Diego State University no pagarán por ningún cuidado, salarios perdidos, ni proporcionarán otra compensación financiera.

Sin embargo, si cree que tiene un reclamo que desea presentar contra State o la Fundación, comuníquese con Asuntos de Posgrado e Investigación – Programa de protección de investigación humana de SDSUal (619) 594-6622 para obtener los formularios de reclamo correspondientes.

<u>Participación Voluntaria</u>: La participación en este estudio es voluntaria. Su elección de participar o no, no influirá en sus relaciones futuras con San Diego State University, la Fundación de San Diego State University, o los Centros de Salud Familiar de San Diego. Si decide participar, puede retirar su consentimiento y detener su participación en cualquier momento sin penalización ni pérdida de los beneficios a los que está autorizado.

<u>Preguntas/Inquietudes:</u> Si tiene alguna pregunta o inquietud sobre la participación en este estudio, por favor pregunte. Si tiene preguntas más adelante sobre la investigación o su participación, puede comunicarse con la investigadora principal, la Dra. Katrina Monroe, PhD, PT (teléfono: 619-594-5553; correo electrónico: ksmonroe@sdsu.edu) o la Dra. Sara Gombatto, PhD, PT (teléfono: 619-594-3288; correo electrónico: sgombatto@sdsu.edu). Si tiene alguna pregunta sobre sus derechos como participante en este estudio, puede comunicarse con un representante del IRB en la División de Asuntos de Investigación de San Diego State University (teléfono: 619-594-6622; correo electrónico: irb@sdsu.edu).

Approved Minimal Risk

Consentimiento para Participar/Derechos del Participante: La Junta de Revisión Institucion Al August 2023 (IRB) de San Diego State University ha aprobado este formulario de consentimiento, como lo indica el sello de la Junta.

Doy mi consentimiento para divulgar mi evaluación relacionada con el estudio y los registros de

| evaluación y tratamiento de fisio<br>garantizar la continuidad de la a | - | y Health Centers of S | San Diego (FHCSD) pa | ara |
|---|---|---|---|---|
| (iniciales del participante | ) | (fecha) | | |
| Doy mi consentimiento para que de fisioterapia y otros registros capacitación. | • | • | | |
| (iniciales del participante | ) | (fech | a) | |
| Doy mi consentimiento para per<br>este estudio se coloquen en un | - | | | <del>;</del> |
| (iniciales del participante | ) | (fecha) | ) | |
| Se le preguntará si está interesa<br>adicionales. Si esta interesado,<br>sobre estos estudios y usted pu<br>independientes de este estudio<br>participando en este estudio. | nos pondremos en<br>ede decidir si partic | contacto con usted p<br>cipar o no en ellos. Es | oor teléfono con inform<br>stos estudios adiciona | les son |
| Doy mi consentimiento de ser codescribe. | ontactado/a para fu | turas oportunidades | de investigación como | se se |
| (iniciales del participante) | | (fecha) | | |
| Su firma a continuación indica que oportunidad de hacer cualquier pestá de acuerdo con participar el su consentimiento para participa de consentimiento. Se le ha dich ninguno de sus derechos legales | oregunta que tenga<br>n el estudio y se le l<br>r en cualquier mom<br>o que al firmar este | sobre el estudio. Su<br>ha dicho que puede o<br>ento. Se le ha dado o | firma también indica q<br>cambiar de opinión y r<br>una copia de este form | etirar<br>nulario |
| Nombre del Participante<br>(letra de imprenta) | Firma del Parti | cipante | Fecha | |
| | Firma del Represe | entante del Proyecto | Fecha | |

Approved Minimal Risk 10 August 2023

## Anexo al Consentimiento para Actuar como Sujeto de Investigación

\_\_\_\_\_ (iniciales del participante) \_\_\_\_\_ (fecha)

incentivo adicional.

| Los investigadores de GOALS/Metas le están reconsiderando en este momento para informarle de un aumento en el incentivo que fue aprobado mediante una enmienda a este proyecto. Marque Si o No abajo para indicar si entiende que está recibiendo este incentivo aparte de la cantidad que ya recibió para mejor reflejar el tiempo que ha dedicado al proyecto. |
|---|
| Yes No |
| Si selecciono Si, coloque sus iniciales y la fecha abajo para reconocer que está de acuerdo con el |

#### Anexo al Consentimiento para Actuar como Sujeto de Investigación

Los investigadores de GOALS/Metas le están reconsiderando en este momento para informarle que información sobre investigaciones adicionales se le presentara en el futuro. Esto fue aprobado mediante una enmienda a este proyecto. Si está interesado, nos pondremos en contacto con usted por teléfono con información sobre estos estudios y usted puede decidir si participar o no en ellos. Estos estudios adicionales son independientes de GOALS/Metas y su decisión sobre ellos no afectarán su capacidad de continuar participando en este estudio.

| Doy mi consentimiento de ser contactado/a para futuras oportunidades de investigación como se describe. |
|---|
| Yes No |
| Si selecciono Si, coloque sus iniciales y la fecha abajo para reconocer que está de acuerdo en se<br>contactado/a para futuras oportunidades de investigación. |
| (iniciales del participante) (fecha) |